CLINICAL TRIAL: NCT02593084
Title: Resistance Training to Optimize Health in Pre-frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAT2015-19
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Frail Elderly
Keywords: Resistance Training; Exercise; Walking; Safety; Feasibility Studies
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher Intensity Resistance Training (Experimental): Participants will take part in a 12-week higher-intensity resistance training protocol.
  Interventions: Behavioral: Higher Intensity Resistance Training
- Lower Intensity Resistance Training (Active Comparator): Participants will take part in a 12-week lower-intensity resistance training protocol that will serve as the active comparator.
  Interventions: Behavioral: Lower Intensity Resistance Training

INTERVENTIONS:
Behavioral: Higher Intensity Resistance Training — Bi-weekly resistance training for 12 weeks using multi-joint movements involving both upper and lower extremities (e.g squats). Participants will perform 3-5 sets of 3-6 repetitions at Rating of Perceived Exertion 8/10. The intervention will be administered by a Physical Therapist or trained fitness professional.
  Other Names: HEaRT
  Arms: Higher Intensity Resistance Training
Behavioral: Lower Intensity Resistance Training — Bi-weekly resistance training for 12 weeks using single-joint movements involving both upper and lower extremities (e.g leg extension). Participants will perform 3-5 sets of 8-10 repetitions at Rating of Perceived Exertion 5/10. The intervention will be administered by a Physical Therapist or trained fitness professional.
  Other Names: LRT
  Arms: Lower Intensity Resistance Training

SUMMARY:
Exercise programs, particularly resistance training programs using weights or resistance bands, can help improve or maintain mobility and function in older adults, preserve independent living, and improve quality of life. This study will examine the safety and feasibility of a novel, higher intensity resistance training program in older adults, and compare the effects with standard care, lower intensity training. It is anticipated that both programs will be safe and feasible, but higher-intensity training will lead to greater improvements in quality of life, mobility and strength, which are part of the physical phenotype definition of frailty and markers of mobility disability.

DETAILED DESCRIPTION:
It is critically important to identify effective strategies to reduce the risk and impact of mobility disability and frailty in older adults. Exercise, particularly resistance training (RT), has the potential to influence a person's ability to navigate around their environment and impact the components of the frailty phenotype which include weakness, physical inactivity, and slowness. Higher training intensities have been used with athletes and younger adults to achieve greater gains in strength, but the feasibility and effectiveness is less established in older persons who exhibit preclinical disability, or are at-risk for mobility decline where conservative protocols are typically employed. Higher intensity RT may be an innovative and effective strategy in preclinical disability pre-frailty to reduce the risk and impact of future frailty and mobility decline.

This study aims to examine: 1) the safety and feasibility of a 12-week higher intensity RT protocol in community dwelling older adults at risk for mobility disability, and 2) the effects of this protocol on walking, balance, muscle strength, quality of life compared to lower intensity RT

It is hypothesized that the higher intensity RT: 1) is safe and feasible for at-risk community-dwelling older adults, 2) more effective in improving walking, balance, muscle strength, and quality of life than lower intensity RT

ELIGIBILITY:
Inclusion Criteria:

* self-reported mobility limitations
* living in the community
* not currently engaged in regular resistance training
* able to follow instructions

Exclusion Criteria:

* contraindications for intensive resistance training (e.g. recent cardiovascular event, fracture within the past 12 months)
* musculoskeletal injuries for which intervention participants are receiving concomitant rehabilitation treatments

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Entire duration of the intervention (12 weeks)
Attendance rate | Entire duration of the intervention (12 weeks)
Attrition rate | Entire duration of the intervention (12 weeks)

SECONDARY OUTCOMES:
Timed Up and Go Test | 0, 12, 20 weeks
Short Physical Performance Battery | 0, 12, 20 weeks
Berg Balance Scale | 0, 12, 20 weeks
Activities-Specific Balance Confidence scale | 0, 12, 20 weeks
Muscle strength | 0, 12, 20 weeks
Short Form-36 | 0, 12, 20 weeks
Caregiver Burden Interview Short Form | 0, 12, 20 weeks
Healthcare Utilization Questionnaires | 0, 12, 20 weeks
Peripheral Quantitative Computed Tomography analysis of muscle and bone quality | 0, 12, 20 weeks
EQ-5D-5L | 0, 12, 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ada Tang, PT PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No